CLINICAL TRIAL: NCT01962545
Title: Optimizing Antithrombotic Care in Patients With AtriaL fibrillatiON and Coronary stEnt (OAC-ALONE) Study
Acronym: OAC-ALONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Satoshi Shizuta (Other)
Collaborators: Research Institute for Production Development (Unknown); Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Satoshi Shizuta, Kyoto University, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C740
Record Dates: First submitted 2013-10-05; First posted 2013-10-14 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: Atrial Fibrillation; Percutaneous coronary intervention; Stent; Anticoagulant therapy; Antiplatelet therapy; Warfarin; NOAC; Aspirin; Clopidogrel
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OAC alone (Experimental): OAC includes warfarin or NOAC. The dose of warfarin should be adjusted with the target international normalized ratio (INR) range of 2.0-3.0 for those <70 years and 1.6-2.6 for those =>70 years, which is recommended in the Japanese guidelines. NOAC includes dabigatran 150mg or 110mg twice daily, rivaroxaban 15mg daily with the reduced dose of 10mg daily, apixaban 5mg twice daily with the reduced dose of 2.5mg twice daily, and edoxaban 60mg daily with the reduced dose of 30mg daily.
  Interventions: Drug: OAC alone
- OAC plus single APT (No Intervention): OAC includes warfarin or NOAC. The dose of warfarin should be adjusted with the target INR range of 2.0-3.0 for those <70 years and 1.6-2.6 for those =>70 years, which is recommended in the Japanese guidelines. NOAC includes dabigatran 150mg or 110mg twice daily, rivaroxaban 15mg daily with the reduced dose of 10mg daily, apixaban 5mg twice daily with the reduced dose of 2.5mg twice daily, and edoxaban 60mg daily with the reduced dose of 30mg daily.
  Single APT includes aspirin or clopidogrel. The dose of aspirin is 81-324mg/day and the dose of clopidogrel is 75mg/day.

INTERVENTIONS:
Drug: OAC alone — Single APT with either aspirin or clopidogrel is discontinued in this arm.
  Arms: OAC alone

SUMMARY:
The purpose of the study is to evaluate non-inferiority of oral anticoagulant (OAC) monotherapy to OAC plus single antiplatelet therapy (APT) in patients with atrial fibrillation (AF) and prior (>12 months) coronary stenting.

DETAILED DESCRIPTION:
It has been reported that 5-10% of patients undergoing percutaneous coronary intervention (PCI) have concomitant AF. Most of those patients have an indication for OAC therapy to prevent stroke or systemic thromboembolism, and also for APT to prevent ischemic cardiac events, particularly myocardial infarction (MI) due to stent thrombosis (ST). However, combined use of OAC and APT is associated with increased risk of major bleeding. Thus, we need to balance the risk for stroke or systemic thromboembolism and coronary events against the risk for bleeding complications.

The AF guidelines of European Society of Cardiology (ESC) published in 2010 recommended vitamin-K antagonist (VKA) monotherapy as life-long antithrombotic therapy after 12 months of combined use of VKA plus APT in AF patients undergoing coronary stenting. Single APT with either aspirin or clopidogrel is the commonly used APT regimen in non-AF patients beyond 1-year after PCI-stenting. No APT coverage after coronary stenting was reported to be associated with increased risk for ST. It has not yet been thoroughly clarified whether VKA monotherapy is equally effective as single APT in the prevention of ST, although several RCTs have shown that VKA was more effective than aspirin for the secondary prevention of ischemic cardiac events in post-MI patients mostly untreated with coronary stent, and recent observational studies have suggested the safety of VKA monotherapy beyond 1-year after PCI-stenting. Nevertheless, there have been no RCTs focusing the safety of VKA monotherapy for AF patients in the chronic phase of PCI-stenting.

Also, because phase-3 RCTs comparing warfarin and non-VKA OAC (NOAC) in the prevention of stroke or systemic embolism in AF patients showed no significant difference in the incidence of MI during follow-up, the consensus document of ESC published in 2014 recommended OAC monotherapy with either VKA or NOAC as life-long antithrombotic therapy beyond 1-year after coronary stenting for AF patients. However, there have been no RCTs or observational studies demonstrating the safety of NOAC alone beyond 1-year after PCI-stenting.

Accordingly, we planned a prospective randomized controlled open label trial comparing OAC alone versus OAC plus single APT in AF patients beyond 1-year after PCI-stenting. AF patients receiving OAC with either warfarin or NOAC in combination with single APT with either aspirin or clopidogrel, who underwent PCI-stenting more than 12 months ago, are eligible for the study. Patients are randomly assigned to OAC alone (intervention arm, discontinuing single APT) or OAC plus single APT (control arm, no change in antithrombotic therapy).

The patient enrollment period is approximately 3 years and follow-up duration is at least 1 year. Therefore, the anticipated mean follow-up duration is approximately 2.5-year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a documented history of AF who underwent PCI with stenting >12 months before enrollment.
2. Patients who are treated with OAC (warfarin or NOAC) and an antiplatelet drug (aspirin or clopidogrel), but not with other antiplatelet drugs including ticlopidine, prasugrel, ticagrelor, and cilostazol.
3. In patients treated with warfarin, the INR value at enrollment should be => 1.6, and agreement on dose adjustment of warfarin with the target INR range of 2.0-3.0 for those <70 years and 1.6-2.6 for those =>70 years, which is recommended in the Japanese guidelines, is necessary before enrollment.
4. Patients 20 years or older.
5. Patients with written informed consent.

Exclusion Criteria:

1. Patients who underwent PCI including balloon angioplasty alone within the past 12 months.
2. Patients in whom OAC is scheduled to be discontinued during the follow-up period.
3. Patients with a past history of ST.
4. Patients with a planned coronary revascularization.
5. Patients with a planned cardiovascular or non-cardiovascular surgery.
6. Patients with expectation of survival less than one year.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is a composite of all-cause death, myocardial infarction, and stroke or systemic embolism. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).

SECONDARY OUTCOMES:
The major secondary endpoint of this study is a composite of all-cause death, myocardial infarction, stroke or systemic embolism, and major bleeding. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
Stent thrombosis. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
  Stent thrombosis.
Myocardial infarction. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
  One of the individual components of the primary endpoint.
Stroke or systemic embolism. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
  One of the individual components of the primary endpoint.
All-cause death. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
  One of the individual components of the primary endpoint.
Major bleeding. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
  One of the individual components of the major secondary endpoint.
Cardiovascular death. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).
Heart failure hospitalization. | Day-0 to the day when the finally enrolled patient complete 1-year follow-up (anticipated mean duration: 2.5-year).

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, M.D., Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Japan

REFERENCES:
- [Derived] Matsumura-Nakano Y, Shizuta S, Komasa A, Morimoto T, Masuda H, Shiomi H, Goto K, Nakai K, Ogawa H, Kobori A, Kono Y, Kaitani K, Suwa S, Aoyama T, Takahashi M, Sasaki Y, Onishi Y, Mano T, Matsuda M, Motooka M, Tomita H, Inoko M, Wakeyama T, Hagiwara N, Tanabe K, Akao M, Miyauchi K, Yajima J, Hanaoka K, Morino Y, Ando K, Furukawa Y, Nakagawa Y, Nakao K, Kozuma K, Kadota K, Kimura K, Kawai K, Ueno T, Okumura K, Kimura T; OAC-ALONE Study Investigators. Open-Label Randomized Trial Comparing Oral Anticoagulation With and Without Single Antiplatelet Therapy in Patients With Atrial Fibrillation and Stable Coronary Artery Disease Beyond 1 Year After Coronary Stent Implantation. Circulation. 2019 Jan 29;139(5):604-616. doi: 10.1161/CIRCULATIONAHA.118.036768. PMID 30586700